CLINICAL TRIAL: NCT06582810
Title: Lidocaine Infusion As A Treatment Modality For Headache Following Non-Traumatic Subarachnoid Hemorrhage: A Prospective, Single-Center, Observational Cohort Study
Brief Title: Lidocaine Infusion Treatment for Subarachnoid Hemorrhage Headaches
Status: Recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Ascension Via Christi Hospitals Wichita, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: RKS20230063; 1856VC (Other: University of Kansas School of Medicine Wichita)
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Subarachnoid; Hemorrhage, Nontraumatic; Headache
Keywords: Nontraumatic Subarachnoid Hemorrhage; Headache; Lidocaine Infusion
MeSH Terms: conditions — Hemorrhage; Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lidocaine infusion: Patients will receive a 100 mg intravenous lidocaine bolus followed by an initial infusion at a rate of 2 mg∙kg -1∙h-1 based on ideal body weight. Lidocaine infusions will continue for a minimum of 1 h post-bolus. If headache numeric pain score decreases at all after initiation of infusion, then the rate will drop to 1 mg∙kg -1∙h-1. If headache numeric pain score starts increasing again, then the rate will return to 2 mg∙kg -1∙h-1, otherwise it will remain at 1 mg∙kg -1∙h-1 for up to 48 h.

SUMMARY:
The goal of this observational study is to evaluate intravenous lidocaine efficacy and safety in treating headache following non-traumatic subarachnoid hemorrhage. Through this prospective analysis, the investigators hope to:

1. show that intravenous lidocaine infusion causes a clinically significant reduction in pain scores in patients with moderate/severe headache pain following non-traumatic subarachnoid hemorrhage;
2. show that intravenous lidocaine infusion is safe in treating headache following non-traumatic subarachnoid hemorrhage;
3. and report vasospasm prevalence in the cohort.

Participants will receive lidocaine infusion as treatment for non-traumatic subarachnoid hemorrhage headache and provide pain scores (on a numeric pain scale) every two hours the patients are awake for a maximum of seven days. Monitoring for vasospasm will occur as part of the patients regular medical care.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years;
* Have a favorable neurological status defined as Hunt and Hess score ≤ 3 (as it accounts for patient awareness);
* Can communicate numeric pain scores;
* Are diagnosed with non-traumatic subarachnoid hemorrhage

Exclusion Criteria:

* The patient is diagnosed with traumatic subarachnoid hemorrhage;
* If the patient is < 18 years of age;
* If numeric pain scores could not be captured for > 3 days of hospitalization;
* If the patient had a prior aneurysm;
* Chronic pain not associated with non-traumatic subarachnoid hemorrhage diagnosis;
* A disability before the stroke (> 2 on modified Rankin Scale score);
* A Hunt and Hess score > 3;
* Contraindications to lidocaine (significant cardiac disease, arrhythmia, seizures, previous allergic reaction to lidocaine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited once a diagnosis of non-traumatic subarachnoid hemorrhage has been confirmed and the patients meet the inclusion criteria for the study. The investigators will exclude incarcerated patients and pregnant women from the study, but the investigators will include patients that cannot consent themselves, as long as the patient meets the inclusion criteria, the investigators can gain consent from the patient's legal guardian/representative, and the patient can report a numeric pain score for the full length of the study (every 2 h the patient is awake for up to 7 days).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Reduction of pain | Benefit should be seen within first 24 h of infusion
  Reduction of pain ≥ 2 points in the numeric pain score after lidocaine infusion treatment. The numeric pain score is a score rating severity of pain from 0 to 10, with higher scores meaning worse pain. The reduction in pain scores indicates a decrease in severity of pain.

OTHER OUTCOMES:
Prevalence of vasospasm | Within the first 7 days participants are receiving treatment
  Observe the prevalence of vasospasm in participants that receive lidocaine infusion

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Salgado, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- Ascension Via Christi St. Francis, Wichita, Kansas, United States